CLINICAL TRIAL: NCT02690545
Title: Phase Ib/II Study of the Administration of T Lymphocytes Expressing the CD30 Chimeric Antigen Receptor (CAR) for Relapsed/Refractory CD30+ Hodgkin's Lymphoma and CD30+ Non-Hodgkin's Lymphoma
Brief Title: Study of CD30 CAR for Relapsed/Refractory CD30+ HL and CD30+ NHL
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC1532-ATL
Record Dates: First submitted 2016-02-10; First posted 2016-02-24 (Estimated); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Lymphoma; Lymphoma, Non-Hodgkin; Immune System Diseases; Immunoproliferative Disorders; Lymphatic Diseases; Lymphoproliferative Disorders; Neoplasms; Neoplasms by Histologic Type
Keywords: CAR T cells; CD30; Lymphoma; T Lymphocytes
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin; Immune System Diseases; Immunoproliferative Disorders; Lymphatic Diseases; Lymphoproliferative Disorders; Neoplasms; Neoplasms by Histologic Type

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ATLCAR.CD30 cells (Experimental): Phase Ib: In adults, and separately, in children, two doses will be investigated 1x10^8 cells/m2 and 2x10^8 cells/m^2. The study team will run two independent dose-escalation sequences, one for adults and another one for children. The study team plans to use the 3+3 design and start with a low dose of 1x10^8 cells/m2. If there are no DLT in first 3 patients, the study team will go up to the dose of 2 x 10^8 cells/m2. If there is toxicity in 1/3 patients in the initial cohort, the study team would expand to enroll up to 6 patients. If there are dose limiting toxicities (DLT) at the dose of 2 x 10^8 cells/m^2, the study team will initially decrease the dose to an intermediate dose of 1.5 x 10^8 cells/m^.
  Phase II: The study team planning to enroll 31 patients to contribute data. Sequential boundary will be used to monitor DLT rate.
  Interventions: Biological: ATLCAR.CD30 cells

INTERVENTIONS:
Biological: ATLCAR.CD30 cells — For Phase Ib, in adults and separately in children, two doses will be investigated: 1x10^8 cells/m^2 and 2x10^8 cells/m^2. Phase II patients will receive the dose level decided upon in Phase I.
  Other Names: CAR.CD30 T cells

SUMMARY:
The body has different ways of fighting infection and disease. No single way seems perfect for fighting cancer. This research study combines two different ways of fighting disease: antibodies and T cells. Antibodies are proteins that protect the body from disease caused by bacteria or toxic substances. Antibodies work by binding those bacteria or substances, which stops them from growing and causing bad effects. T cells, also called T lymphocytes, are special infection-fighting blood cells that can kill other cells, including tumor cells or cells that are infected. Both antibodies and T cells have been used to treat patients with cancers. They both have shown promise, but neither alone has been sufficient to cure most patients. This study is designed to combine both T cells and antibodies to create a more effective treatment called autologous T lymphocyte chimeric antigen receptor cells targeted against the CD30 antigen (ATLCAR.CD30) administration.

In previous studies, it has been shown that a new gene can be put into T cells that will increase their ability to recognize and kill cancer cells. The new gene that is put in the T cells in this study makes an antibody called anti-CD30. This antibody sticks to lymphoma cells because of a substance on the outside of the cells called CD30. Anti-CD30 antibodies have been used to treat people with lymphoma, but have not been strong enough to cure most patients. For this study, the anti-CD30 antibody has been changed so that instead of floating free in the blood it is now joined to the T cells. When an antibody is joined to a T cell in this way it is called a chimeric receptor. These CD30 chimeric (combination) receptor-activated T cells seem to kill some of the tumor, but they do not last very long in the body and so their chances of fighting the cancer are unknown.

The purpose of this research study is to establish a safe dose of ATLCAR.CD30 cells to infuse after lymphodepleting chemotherapy and to estimate the number patients whose cancer does not progress for two years after ATLCAR.CD30 administration. This study will also look at other effects of ATLCAR.CD30 cells, including their effect on the patient's cancer.

DETAILED DESCRIPTION:
STUDY OBJECTIVES

Primary Objective (Phase Ib portion of Study) To establish a safe dose (ie, number cells/m2) of ATLCAR.CD30 to infuse after lymphodepletion with bendamustine in adult patients with CD30+ refractory/relapsed Hodgkin lymphoma (HL) and non-Hodgkin lymphoma (NHL).

To establish a safe dose (ie, number cells/m2) of ATLCAR.CD30 to infuse after lymphodepletion with bendamustine and fludarabine in pediatric patients with CD30+ refractory/relapsed Hodgkin lymphoma (HL) and non-Hodgkin lymphoma (NHL).

Primary Objective (Phase II portion of study) To estimate 2 year progression free survival (PFS) after administration of ATLCAR.CD30 in combined adult/pediatric patients with CD30+ refractory/relapsed HL and NHL

Secondary Objectives

To estimate 2 year overall survival (OS) after administration of CAR.CD30 transduced ATL following lymphodepletion with bendamustine in adult patients with CD30+ relapsed/refractory HL and NHL.

To estimate 2 year OS after administration of CAR.CD30 transduced ATL following lymphodepletion with bendamustine and fludarabine in adult and pediatric patients with CD30+ relapsed/refractory HL and NHL.

To estimate 2 year PFS after administration of ATLCAR.CD30 following lymphodepletion with bendamustine in adult patients with CD30+ refractory/relapsed HL and NHL.

To estimate 2 year PFS after administration of ATLCAR.CD30 following lymphodepletion with bendamustine and fludarabine in adult and pediatric patients with CD30+ refractory/relapsed HL and NHL.

To estimate the objective response rate as defined by the Lugano Classification78 for CAR.CD30 transduced ATL following lymphodepletion with bendamustine when administered in adult patients with CD30+ relapsed/refractory HL and NHL.

To estimate the objective response rate as defined by the Lugano Classification78 for CAR.CD30 transduced ATL following lymphodepletion with bendamustine and fludarabine when administered in adult and pediatric patients with CD30+ relapsed/refractory HL and NHL.

To estimate duration of response after administration of CAR.CD30 transduced ATL following lymphodepletion with bendamustine in adult patients with CD30+ relapsed/refractory HL and NHL

To estimate duration of response after administration of CAR.CD30 transduced ATL following lymphodepletion with bendamustine and fludarabine in adult and pediatric patients with CD30+ relapsed/refractory HL and NHL

To further describe the adverse events associated with CAR.CD30 transduced ATL when administered in adult and pediatric patients with CD30+ relapsed/refractory HL and NHL.

To evaluate the safety of bendamustine alone or combined with fludarabine as lymphodepleting agents prior to infusion of CAR.CD30 transduced ATL in adult patients.

To evaluate the safety of bendamustine and fludarabine as lymphodepleting agents prior to infusion of CAR.CD30 transduced ATLs in pediatric patients.

To measure the survival of ATLCAR.CD30 in vivo when infused after lymphodepletion with bendamustine.

To measure the survival of ATLCAR.CD30 in vivo when infused after lymphodepletion with bendamustine and fludarabine.

To measure patient-reported symptom, physical function, and health-related quality of life at baseline and over time in adult patients treated with CAR.CD30 T cells.

Primary Endpoint (Phase Ib)

Toxicity will be classified and graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, version 4.0) and Cytokine Release Syndrome (CRS) toxicity will be graded according to the CRS Management Guidelines and CRS Toxicity Grading Scale

Primary Endpoint (Phase II)

PFS is defined from day of ATLCAR.CD30 infusion to relapse (in patients with a documented complete response at time of cell infusion) or progression (in patients without complete response at time of cell infusion), or death as a result of any cause per the Lugano classification

Secondary Endpoints

Overall survival will be measured from the date of administration of CAR.CD30 transduced ATL to date of death and will be measured separately in subjects receiving bendamustine alone for lymphodepletion and those receiving a combination of bendamustine and fludarabine for lymphodepletion.

Progression free survival is defined from day of ATLCAR.CD30 infusion to relapse (in patients with a documented complete response at time of cell infusion) or progression (in patients without complete response at time of cell infusion), or death as a result of any cause per the Lugano classification78 and will be measured separately in subjects receiving bendamustine alone for lymphodepletion and those receiving a combination of bendamustine and fludarabine for lymphodepletion.

The objective response rate will be defined as the rate of complete responses (CR) + partial responses (PR) as determined by the Lugano classification78 and will be measured separately in subjects receiving bendamustine alone for lymphodepletion and those receiving a combination of bendamustine and fludarabine for lymphodepletion.

The duration of response will be defined as time from documentation of tumor response to disease progression and will be measured separately in subjects receiving bendamustine alone for lymphodepletion and those receiving a combination of bendamustine and fludarabine for lymphodepletion.

Toxicity will be classified and graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, version 4.0). S

Persistence of CAR.CD30 T cells in vivo will be determined by quantitative PCR and flow cytometry in peripheral blood samples and will be measured separately in subjects receiving bendamustine alone for lymphodepletion and those receiving a combination of bendamustine and fludarabine for lymphodepletion.

For adult patients: Patient reported symptoms will be measured using selected symptoms from the NCI PRO-CTCAE. Patient-reported physical function will be measured using the PROMIS Physical Function Score derived from the PROMIS Physical Function Short Form 20a v1.0. Patient-reported health-related quality of life will be measured using the PROMIS Global Health Score derived from the PROMIS Global Health Short Form v1.0-1.1.

OUTLINE

Cell Procurement

Up to 100 mL per collection (up to 3 collections) of peripheral blood will be obtained from patients for cell procurement. In patients with low (CD3 count as assayed by flow cytometry less than 200/μl) T-cell count in the peripheral blood, a leukopheresis may be performed to isolate sufficient T cells. The parameters for pheresis will be 2 blood volumes.

ATLCAR.CD30 Cells Administration

ATLCAR.CD30 cells will be administered as described below 1-14 days (preferably 1-2 days) after lymphodepletion with bendamustine and fludarabine. ATLCAR.CD30 cells will be given by a licensed provider (oncology nurse or physician) via intravenous injection over 1-10 minutes through either a peripheral or a central line. The expected volume will be 1-50cc. Patients with a partial response or stable disease at 6 weeks may receive a second infusion of ATLCAR.CD30 if cells are available. Note: Lymphodepletion with bendamustine and fludarabine will occur for three consecutive days and may be given prior to a second infusion of cells (if applicable).

Duration of Therapy

Therapy in Lineberger Comprehensive Cancer Center (LCCC) 1532 involves 1-2 infusions of ATLCAR.CD30 cells. Treatment with one infusion will be administered unless:

* Patient decides to withdraw from study treatment, OR
* General or specific changes in the patient's condition render the patient unacceptable for further treatment in the judgment of the investigator.

Duration of Follow-up

Patients will be followed for up to 15 years for Replication Competent Retrovirus (RCR) evaluation or until death, whichever occurs first. Patients removed from study for unacceptable adverse events will be followed until resolution or stabilization of the adverse event.

ELIGIBILITY:
Inclusion Criteria Prior to Cell Procurement

Informed consent explained to, understood by and signed by the subject or legal guardian for pediatric subjects; subject and/or legal guradian given a copy of informed consent form for procurement

Ages 3 to 17 years of age for pediatric subjects (weight must be ≥10kg), and for adults ages ≥18 years of age

Diagnosis of recurrent HL or NHL in subjects who have failed >2 prior treatment regimens. Subjects relapsed after autologous or allogeneic stem cell transplant are eligible for this study.

CD30+ disease (result can be pending at the time of cell procurement, but must be confirmed prior to treatment with ATLCAR.CD30 cells). NOTE: CD30+ disease requires documented CD30 expression by immunohistochemistry based on the institutional hematopathology standard.

Karnofsky or Lansky score of >60% (Karnofsky for ≥16 years old and Lansky for <16 years old)

Evidence of adequate organ function as defined by:

* Hemoglobin ≥ 8.0 g/dL (transfusion independent for 2 weeks prior to enrollment)
* Total bilirubin ≤ 1.5 × ULN, unless attributed to Gilbert's Syndrome
* AST ≤ 3 × ULN
* Serum creatinine ≤ 1.5 × ULN
* For subjects <18 years old use the following table for serum creatinine requirements:

Maximum Serum Creatinine (mg/dL) Age (years) Male Female 3 to <6 ≤0.8 ≤0.8 6 to <10 ≤1.0 ≤1.0 10 to <13 ≤1.2 ≤1.2 13 to <16 ≤1.5 ≤1.4 ≥16 and <18 ≤1.7 ≤1.4

Negative serum pregnancy test in females within 72 hours prior to procurement or documentation that the subject is post-menopausal or premenarchal.

Women of childbearing potential (WOCBP) should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study, and for 6 months after the study is concluded. WOCBP are those who have not been surgically sterilized or have not been free from menses for >1 year.

• Postmenopausal status must be confirmed with documentation of absence of menses for >1 year.

Exclusion Criteria Prior to Cell Procurement

Pregnant or lactating

Tumor in a location where enlargement could cause airway obstruction

Must not have an Active infection with human immunodeficiency virus (HIV), Hepatitis B Virus (HBV))or, Hepatitis C virus (HCV) (can be pending at the time of cell procurement; only subjects meeting the criteria as so described will be infused). Note: To meet eligibility subjects are required to have negative HIV antibody, negative for Hepatitis B surface antigen and negative for HCV antibody or viral load.

Inclusion Criteria Prior to Lymphodepletion

Informed consent explained to, understood by and signed by the subject or legal guardian for pediatric subjects; subject and/or legal guradian given a copy of informed consent form.

CD30+ disease (result can be pending at the time of cell procurement, but must be confirmed prior to lymphodepletion); Note: CD30+ disease requires documented CD30 expression by immunohistochemistry based on the institutional hematopathology standard.

Prior to administration of lymphodepletion:

* Absolute neutrophil count (ANC) is > 1.0 × 10^9/L
* Platelet count > 75 × 10^9/L
* For Grade 4 neutropenia, Grade ≥3 febrile neutropenia, or Grade 4 thrombocytopenia, hold bendamustine until toxicity resolve to Grade ≤2

For WOCBP negative serum pregnancy test within 72 hours prior to lymphodepletion.

Imaging results from within 7 days (30 days in subjects with cutaneous T cell lymphoma) prior to lymphodepletion. Subjects who have received bridging chemotherapy must have imaging performed at least 3 weeks after most recent therapy (imaging does not need to be repeated if it is within 7 days prior to lymphodepletion).

Karnofsky or Lansky score of >60% (Karnofsky for pediatric subjects ≥16 years old and Lansky for <16 years old).

Available autologous transduced activated T cells that meet the Certificate of Analysis (CofA) acceptance criteria.

Women of childbearing potential (WOCBP) should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study, and for 6 months after the study is concluded. WOCBP are those who have not been surgically sterilized or have not been free from menses for > 1 year.

Exclusion Criteria Prior to Lymphodepletion

Received any investigational agents or received any tumor vaccines within the previous six weeks prior to cell infusion.

Received anti-CD30 antibody-based therapy within the previous 4 weeks prior to cell infusion.

Received chemotherapy within the previous 3 weeks prior to lymphodepletion.

Subject has rapidly progressive disease, per treating oncologist's discretion.

Subject is not a good candidate for CAR T cell therapy, per treating oncologist's discretion.

Pregnant or lactating.

Tumor in a location where enlargement could cause airway obstruction.

Current use of systemic corticosteroids at doses equivalent of ≥10mg prednisone daily or its equivalent; those receiving <10mg daily may be enrolled at discretion of investigator. Inhaled steroids are allowed.

For pediatric subjects, physiologic replacement hydrocortisone at doses 6-12 mg/m2/day is allowed. Equivalently dosed alternative steroids are allowed at discretion of investigator, though not to exceed 10mg prednisone per day. Inhaled steroids are allowed.

Subjects on strong inhibitors of CYP1A2 (e.g., fluvoxamine, ciprofloxacin) as these may increase plasma concentrations of bendamustine, and decrease plasma concentrations of its metabolites. See http://medicine.iupui.edu/clinpharm/ddis/ for an updated list of strong inhibitors of CYP1A2. Details are given in the protocol.(This applies to subjects who receive bendamustine for lymphodepletion (required) up through 72 hours after the last dose of bendamustine.)

Active infection with HIV, HBV or HCV (can be pending at the time of cell procurement; only subjects meeting the criteria as so described will be infused. Subjects are required to have negative HIV antibody or negative for Hepatitis B surface antigen and negative HCV antibody or viral load.

Hepatitis B: Subjects who are positive for Hepatitis B Surface Antigen are excluded. Subjects who are Hepatitis B Surface Antigen negative but hepatitis B core Antibody positive must have their hepatitis B viral load checked. These subjects will be excluded if their viral load is positive at baseline. Subjects who are core antibody positive and viral load negative at baseline will be considered eligible if the subject has initiated an anti-HBV prophylaxis regimen prior to lymphodepletion.

Inclusion Criteria Prior to Infusion of ATLCAR.CD30 Cells

Evidence of adequate organ function as defined by:

* Total bilirubin ≤1.5 × ULN, unless attributed to Gilbert's Syndrome
* AST ≤3 × ULN
* Serum creatinine ≤1.5 × ULN
* Pulse oximetry of >90% on room air
* For subjects <18 years old use following table for serum creatinine requirements:

Maximum Serum Creatinine (mg/dL) Age (years) Male Female 3 to <6 ≤0.8 ≤0.8 6 to <10 ≤1.0 ≤1.0 10 to <13 ≤1.2 ≤1.2 13 to <16 ≤1.5 ≤1.4 ≥16 and <18 ≤1.7 ≤1.4

Karnofsky or Lansky score of >60% (Karnofsky for ≥16 years old and Lansky for <16 years old)

Available autologous transduced activated T cells that meet the Certificate of Analysis (CofA) acceptance criteria.

Women of childbearing potential (WOCBP) should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study, and for 6 months after the study is concluded. WOCBP are those who have not been surgically sterilized or have not been free from menses for > 1 year.

Exclusion Criteria Prior to Infusion of ATLCAR.CD30 Cells

Received any investigational agents or received any tumor vaccines within the previous six weeks prior to cell infusion.

Received anti-CD30 antibody-based therapy within the previous 4 weeks prior to cell infusion.

Tumor in a location where enlargement could cause airway obstruction.

Subject has rapidly progressive disease, per treating oncologist's discretion.

Subject is not a good candidate for CAR T cell therapy, per treating oncologist's discretion.

Current use of systemic corticosteroids at doses ≥10 mg prednisone daily or its equivalent; those receiving <10 mg daily may be enrolled at discretion of investigator. Inhaled steroids are allowed For pediatric subjects, physiologic replacement hydrocortisone at doses 6-12mg/m2/day is allowed. Equivalently dosed alternative steroids are allowed at discretion of investigator, though not to exceed 10mg prednisone per day. Inhaled steroids are allowed.

Active infection with HIV or HCV (can be pending at the time of cell procurement; only subjects meeting the criteria as so described will be infused). Subjects are required to be negative for HIV and negative for Hepatitis B surface antigen, and negative HCV antibody or viral load.

Hepatitis B: Subjects who are positive for Hepatitis B Surface Antigen are excluded. Subjects who are Hepatitis B Surface Antigen negative but hepatitis B core antibody positive must have their hepatitis B viral load checked. These subjects will be excluded if their viral load is positive at baseline. Subjects who are core antibody positive and viral load negative at baseline will be considered eligible. These subjects must be receiving antiviral prophylaxis initiated prior to lymphodepletion.

Eligibility Criteria Prior to Lymphodepletion for Second Infusion (Optional) Note: Subjects may receive a second infusion without prior lymphodepletion if they meet the eligibility criteria at the time of infusion, but do not meet the eligibility requirements for adequate bone marrow function and platelet counts.

Karnofsky or Lansky score of >60% (Karnofsky for ≥16 years old and Lansky for <16 years old).

WOCBP must be willing to use 2 methods of birth control or be surgically sterile , or abstain from heterosexual activity for the course of the study, or for 6 months after the study is concluded. WOCBP are those who have not been surgically sterilized or have not been free from menses for > 1 year.

Subject must not be pregnant or lactating within 7 days of infusion.

Must not have tumor in a location where enlargement could cause airway obstruction.

Subjects must have imaging results confirming active disease from within 30 days prior to lymphodepletion with the exception of cutaneous lymphoma subjects who do not need to repeat scans prior to the second cell infusion if the baseline scans showed lymph nodes ≤ 1.5cm at baseline.

Must not have current use of systemic corticosteroids at doses ≥10 mg prednisone daily or its equivalent; those receiving <10mg daily may be enrolled at discretion of the Investigator

Evidence of adequate organ function as defined by:

* ANC>1.0 × 10^9/L
* Platelets >75 × 10^9/L
* Total bilirubin ≤1.5 × ULN, unless attributed to Gilbert's syndrome
* AST ≤3 × ULN
* Serum creatinine ≤1.5 × ULN
* Pulse oximetry of > 90% on room air
* For subjects <18 years old use following table for serum creatinine requirements:

Maximum Serum Creatinine (mg/dL) Age (years) Male Female 3 to <6 ≤0.8 ≤0.8 6 to <10 ≤1.0 ≤1.0 10 to <13 ≤1.2 ≤1.2 13 to <16 ≤1.5 ≤1.4 ≥16 and <18 ≤1.7 ≤1.4

Negative serum pregnancy test within 72 hours prior to lymphodepletion or documentation that the subject is post-menopausal. Post-menopausal status must be confirmed with documentation of absence of menses for > 1 year or documentation of surgical menopause involving bilateral oophorectomy.

Subject cannot be on strong inhibitors of CYP1A2 (e.g., fluvoxamine, ciprofloxacin) as these may increase plasma concentrations of bendamustine, and decrease plasma concentrations of its metabolites. See http://medicine.iupui.edu/clinpharm/ddis/ for an updated list of strong inhibitors of CYP1A2. (This applies to subjects who receive bendamustine for lymphodepletion (required) up through 72 hours after the last dose of bendamustine)

Subject is a good candidate for treatment with ATLCAR.CD30 per the investigator's discretion.

Eligibility Criteria Prior to Second Infusion (Optional)

No evidence of uncontrolled infection or sepsis.

Subject must not have undergone bridging chemotherapy (or other anti-cancer therapies, which are not mandated by the protocol) prior to the second infusion.

Evidence of adequate organ function as defined by:

* Total bilirubin ≤2 × ULN, unless attributed to Gilbert's syndrome
* AST ≤3 × ULN
* ALT ≤3 × ULN
* Serum creatinine ≤1.5 × ULN
* Pulse oximetry of >90% on room air
* For subjects <18 years old use following table for serum creatinine requirements:

Maximum Serum Creatinine (mg/dL) Age (years) Male Female 3 to <6 ≤0.8 ≤0.8 6 to <10 ≤1.0 ≤1.0 10 to <13 ≤1.2 ≤1.2 13 to <16 ≤1.5 ≤1.4

≥16 and <18 ≤1.7 ≤1.4

Subject has no clinical indication of rapidly progressing disease in the opinion of the treating physician

Subject is a good candidate for treatment with ATLCAR.CD30 per the investigator's discretion.

If subjects have had positive hepatitis B core antibody testing at baseline, they must not have had re-activation of the Hepatitis B virus since baseline testing.

Subject must not be pregnant or lactating within 7 days of infusion.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-08-26 (Actual); Primary Completion 2025-12-16 (Actual); Study Completion 2039-11-04 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability of ATLCAR.CD30 cells to establish a safe dose after lymphodepletion with bendamustine in adult patients | 6 weeks
  Toxicity will be classified and graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, version 4.0). Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living (ADL). Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE
Number of participants with adverse events as a measure of safety and tolerability of ATLCAR.CD30 cells to establish a safe dose after lymphodepletion after lymphodepletion with bendamustine and fludarabine in pediatric patients | 6 weeks
  Toxicity will be classified and graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, version 4.0). Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living (ADL). Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE
2 year progression free survival (PFS) after administration of ATLCAR.CD30 in combined adult/pediatric patients with CD30+ refractory/relapsed HL and NHL. | 2 years
  PFS is defined from day of ATLCAR.CD30 infusion to relapse (in patients with a documented complete response at time of cell infusion) or progression (in patients without complete response at time of cell infusion), or death as a results of any cause per the Lugano classification.

SECONDARY OUTCOMES:
2 year overall survival (OS) after administration of CAR.CD30 transduced ATL following lymphodepletion with bendamustine and fludarabine in adult and pediatric patients with CD30+ relapsed/refractory HL and NHL. | 2 years
  Overall survival will be measured from the date of administration of CAR.CD30 transduced ATL to the date of death and will be measured in subjects receiving a combination of bendamustine and fludarabine for lymphodepletion.
2 year overall survival (OS) after administration of ATLCAR.CD30 transduced ATl following lymphodepletion with bendamustine in adult patients with CD30+ refractory/relapsed HL and NHL | 2 years
  Overall survival will be measured from the date of administration of CAR.CD30 transduced ATL to date of death and will be measured in subjects receiving bendamustine alone.
2 year progression free survival after administration of ATLCAR.CD30 following lymphodepletion with bendamustine in adult patients with CD30+ in adult patients with CD30+ refractory/relapsed HL and NHL. | 2 years
  Progression free survival is defined from day of ATLCAR.CD30 infusion to relapse (in patients with a documented complete response at time of cell infusion) or progression (in patients without complete response at time of cell infusion), or death as a result of any cause per the Lugano classification and will be measured in subjects receiving bendamustine alone.
2 year progression free survival after administration of ATLCAR.CD30 following lymphodepletion with bendamustine and fludarabine in adult and pediatric patients with CD30+ refractory/relapsed HL and NHL. | 2 years
  Progression free survival is defined from day of ATLCAR.CD30 infusion to relapse (in patients with a documented complete response at time of cell infusion) or progression (in patients without complete response at time of cell infusion), or death as a result of any cause per the Lugano classification and will be measured in subjects receiving a combination of bendamustine and fludarabine for lymphodepletion.
Objective response rate as defined by the Lugano Classification for CAR.CD30 transduced ATL following lymphodepletion with bendamustine when administered in adult patients with CD30+ relapsed/refractory HL and NHL | 6 weeks
  The objective response rate will be defined as the rate of complete responses (CR) + partial responses (PR) as determined by the Lugano classification and will be measured in subjects receiving bendamustine alone for lymphodepletion.
Objective response rate as defined by the Lugano classification for CAR.CD30 transduced ATL following lymphodepletion with bendamustine and fludarabine when administered in adult and pediatric patients with CD30+ relapsed/refractory HL and NHL. | 6 weeks
  The objective response rate will be defined as the rate of complete responses (CR) + partial responses (PR) as determined by the Lugano classification and will be measured in subjects receiving bendamustine and fludarabine for lymphodepletion.
Duration of response after administration of CAR.CD30 transduced ATL following lymphodepletion with bendamustine in adult patients with CD30+ relapsed/refractory HL and NHL. | 15 years
  Duration of response will be defined as time from documentation of tumor response to disease progression and will be measured in subjects receiving bendamustine alone for lymphodepletion.
Duration of response after administration of CAR.CD30 transduced ATL following lymphodepletion with bendamustine and fludarabine in adult and pediatric patients with CD30+ relapsed/refractory HL and NHL. | 15 years
  Duration of response will be defined as time from documentation of tumor response to disease progression and will be measured in subjects receiving a combination of bendamustine and fludarabine for lymphodepletion.
Adverse events associated with CAR.CD30 transduced ATL when administered in adult and pediatric patients with CD30+ relapsed/refractory HL and NHL. | 6 weeks
  Toxicity will be classified and graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, version 4.0).
Number of participants with adverse events as a measure of safety and tolerability of bendamustine and fludarabine as lymphodepleting agents | 6 weeks
  Toxicity will be classified and graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, version 4.0).
Number of adverse events as a measure of safety and tolerability of bendamustine and fludarabine as lymphodepleting agents prior to infusion of CAR.CD30 transduced ATLs in pediatric patients. | 6 weeks
  Toxicity will be classified and graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, version 4.0).
Survival of ATLCAR.CD30 in vivo when infused after lymphodepletion with bendamustine. | 15 years
  Persistence of CAR.CD30 T cells in vivo will be determined by quantitative PCR and flow cytometry in peripheral blood samples and will be measured in subjects receiving bendamustine alone for lymphodepletion.
To measure the survival of ATLCAR.CD30 in vivo when infused after lymphodepletion with bendamustine and fludarabine. | 15 years
  Persistence of CAR.CD30 T cells in vivo will be determined by quantitative PCR and flow cytometry in peripheral blood samples and will be measured in subjects receiving bendamustine in combination with fludarabine for lymphodepletion
Measure patient-reported symptoms using selected symptom items from the NCI Patient Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE) at baseline and over time in adult patients treated with CAR.CD30 T cells. | 15 years
  The NCI Patient Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE) is a patient-reported outcome measurement system developed to characterize the frequency, severity and interference of 78 symptomatic treatment toxicities. Each item is scored from 0 to four.
Measure patient-reported quality of life using the PROMIS Global Health (PROMIS GHS SF v1.0-1.1) at baseline and over time in adult patients treated with CAR.CD30 T cells. | 15 years
  The PROMIS Global Health Short Form is a 10-item instrument representing multiple domains relating to overall health. Each item has a scale from 1 (poor) to 5 (excellent). Item 7, 8, and 10 are recoded. The global physical health score is generated by summing responses to Global03, Global06, Global07 rescored, Global08 rescored. The Global Mental Health score is generated by summing responses to Global02, Global04, Global05, Global10 Rescored.
Measure patient reported quality of life using the PROMIS Physical Function (PROMIS Physical Function SF20a) at baseline and over time in adult patients treated with CAR.CD30 T cells. | 15 years
  The PROMIS Physical Function short form is a 20 item instrument that measures self-reported capability rather than actual performance of physical activities. This includes the functioning of one's upper extremities (dexterity), lower extremities (walking or mobility), and central regions (neck, back), as well as instrumental activities of daily living, such as running errands. Each item has five response options ranging in value from 1 (unable to do) to 5 (without any difficulty). To items are summed to find the overall raw score.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Beaven, MD, Principal Investigator — Director, UNC Lineberger Lymphoma Program
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tschernia NP, Heiling H, Deal AM, Cheng C, Babinec C, Gonzalez M, Morrison JK, Dittus C, Dotti G, Beaven AW, Serody JS, Wood WA, Savoldo B, Grover NS. Patient-reported outcomes in CD30-directed CAR-T cells against relapsed/refractory CD30+ lymphomas. J Immunother Cancer. 2023 Aug;11(8):e006959. doi: 10.1136/jitc-2023-006959. PMID 37527906
- [Derived] Voorhees TJ, Zhao B, Oldan J, Hucks G, Khandani A, Dittus C, Smith J, Morrison JK, Cheng CJ, Ivanova A, Park S, Shea TC, Beaven AW, Dotti G, Serody J, Savoldo B, Grover N. Pretherapy metabolic tumor volume is associated with response to CD30 CAR T cells in Hodgkin lymphoma. Blood Adv. 2022 Feb 22;6(4):1255-1263. doi: 10.1182/bloodadvances.2021005385. PMID 34666347
- [Derived] Ramos CA, Grover NS, Beaven AW, Lulla PD, Wu MF, Ivanova A, Wang T, Shea TC, Rooney CM, Dittus C, Park SI, Gee AP, Eldridge PW, McKay KL, Mehta B, Cheng CJ, Buchanan FB, Grilley BJ, Morrison K, Brenner MK, Serody JS, Dotti G, Heslop HE, Savoldo B. Anti-CD30 CAR-T Cell Therapy in Relapsed and Refractory Hodgkin Lymphoma. J Clin Oncol. 2020 Nov 10;38(32):3794-3804. doi: 10.1200/JCO.20.01342. Epub 2020 Jul 23. PMID 32701411
- See also: University of North Carolina (UNC) Lineberger Comprehensive Cancer Center — http://unclineberger.org